CLINICAL TRIAL: NCT00092768
Title: A 26-Week, Randomized, Placebo- and Active-Comparator-Controlled, Parallel-Group, Double-Blind, 2-Part Study to Assess the Safety and Efficacy of Etoricoxib 30 mg Versus Celecoxib 200 mg in Patients With Osteoarthritis (Study 1)
Brief Title: A Study of MK0663 and an Approved Drug in the Treatment of Osteoarthritis (0663-076)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-076; 2004_057
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Arcoxia
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib
Drug: Comparator: celecoxib

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of an investigational drug and an approved drug in the treatment of osteoarthritis of the knee and hip.

DETAILED DESCRIPTION:
The duration of treatment is 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee or hip which requires treatment with a medication to obtain pain relief

Exclusion Criteria:

* Any known allergy to the study drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2005-02-01 (Actual); Study Completion 2005-02-01 (Actual)

PRIMARY OUTCOMES:
Osteoarthritis of the knee & hip as assessed by WOMAC VA 3.0 pain and physical function subscales, Patient/Investigator assessments of disease and response to therapy over 12 weeks of treatment.

SECONDARY OUTCOMES:
Maintenance of clinical efficacy as assessed by WOMAC subscales and Patient assessments over a 26-wks of treatment. Safety / tolerability over a 12-wk and 6-mo treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Bingham CO 3rd, Sebba AI, Rubin BR, Ruoff GE, Kremer J, Bird S, Smugar SS, Fitzgerald BJ, O'Brien K, Tershakovec AM. Efficacy and safety of etoricoxib 30 mg and celecoxib 200 mg in the treatment of osteoarthritis in two identically designed, randomized, placebo-controlled, non-inferiority studies. Rheumatology (Oxford). 2007 Mar;46(3):496-507. doi: 10.1093/rheumatology/kel296. Epub 2006 Aug 27. PMID 16936327
- [Background] Bingham CO 3rd, Bird SR, Smugar SS, Xu X, Tershakovec AM. Responder analysis and correlation of outcome measures: pooled results from two identical studies comparing etoricoxib, celecoxib, and placebo in osteoarthritis. Osteoarthritis Cartilage. 2008 Nov;16(11):1289-93. doi: 10.1016/j.joca.2008.04.009. Epub 2008 Jun 2. PMID 18514551
- [Background] Bingham CO 3rd, Smugar SS, Wang H, Tershakovec AM. Early response to COX-2 inhibitors as a predictor of overall response in osteoarthritis: pooled results from two identical trials comparing etoricoxib, celecoxib and placebo. Rheumatology (Oxford). 2009 Sep;48(9):1122-7. doi: 10.1093/rheumatology/kep184. Epub 2009 Jul 9. PMID 19589894